CLINICAL TRIAL: NCT05716516
Title: Phase II Study of Estradiol Therapy to Target ER-Mutant and ER-Wild-Type ER+ Metastatic or Advanced Breast Cancer
Brief Title: STUDY02001740;22SCH740: Estradiol For ER+ Advanced Breast Cancer (ESTHER)
Acronym: ESTHER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Muhammad.Z.Afzal, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001740; NCI-2023-05453 (Other: National Cancer Institute)
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic; Locally advanced; Estradiol therapy; Estrogen therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Other): Treatment Phase: Patients will be treated with 17b-estradiol until disease progression. At this point, the patient will end protocol therapy
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Estradiol is a therapeutic option for the treatment of advanced ER+ breast cancer
  Other Names: Estrace

SUMMARY:
Determine whether subjects harboring ESR1-mutant/amplified breast cancer have a higher rate of clinical benefit from 17b-estradiol therapy than subjects with ESR1-wild-type breast cancer

DETAILED DESCRIPTION:
Patients with endocrine-resistant breast cancer are eligible. Treatment Phase: Patients will be treated with 17b-estradiol until disease progression. At this point, the patient will end protocol therapy. Clinical benefit, progression-free survival, objective response, tumor metabolic response, and toxicity will be determined. Observational Phase (optional): After disease progression on 17b-estradiol, patients will be treated at their oncologist's discretion. Clinical benefit, progression-free survival, and objective response will be measured during this line of treatment of physician's choice until another instance of disease progression. In consented subjects who undergo a clinically indicated tumor biopsy of recurrent or metastatic disease prior to the start of 17b-estradiol treatment, when feasible, acquisition of additional tumor tissue is requested for research purposes. Optional: patients will be asked to provide tumor tissue via a research biopsy on Day 3-4 of 17b-estradiol treatment. Archived tumor tissue and clinical-grade tumor and plasma DNA/RNA sequencing results will be used for research purposes. Blood samples will be obtained at baseline, on Day 3-4 of 17b-estradiol therapy (optional), and upon disease progression on 17b-estradiol. Plasma and buffy coat will be extracted and frozen. Tumor tissue and plasma specimens will be analyzed to identify molecular biomarkers predictive of sensitivity/resistance to 17b-estradiol therapy

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with ER+ breast cancer.
* Metastatic or locoregional recurrence not amenable to treatment with curative
* intent.
* Received ≥1 prior line of endocrine-based therapy (e.g., including tamoxifen, aromatase inhibitors, fulvestrant, or combinations) in the advanced/metastatic setting

Exclusion Criteria:

* During the study Treatment Phase with 17b-estradiol, no concurrent anti-cancer therapies are allowed with the following exceptions:

  * Exception: Trastuzumab is allowed for the treatment of subjects with a history of HER2+ disease, and will be used at the physician's discretion.
  * Exception: Anti-resorptive bone therapies (e.g., bisphosphonates, denosumab) are permitted.
* Any investigational cancer therapy in the last 3 weeks.
* Known CNS disease, unless clinically stable for ≥ 3 months.
* History of any of the following:

  * Deep venous thrombosis.
  * Pulmonary embolism.
  * Stroke.
  * Acute myocardial infarction.
  * Congestive heart failure.
  * Previous malignancy not treated with curative intent, or with an estimated recurrence risk ≥30%.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate | 12 months
  The clinical benefit rate (complete responses + partial responses + stable disease at 24 weeks) will be ascertained and compared between subjects treated with 17b-estradiol harboring amplified/mutant ESR1 and wild-type ESR1.

SECONDARY OUTCOMES:
Objective response rate | 8 weeks
  The objective response rate (complete + partial responses) to the first 8 weeks of treatment with 17b-estradiol will be ascertained and compared between subjects harboring amplified/mutant ESR1 and wild-type ESR1.
Progression-free survival | 12 months
  Progression-free survival with 17b-estradiol treatment will be ascertained and compared between subjects harboring amplified/mutant ESR1 and wild-type ESR1.
Tumor Metabolic response | 12 months
  Tumor metabolic response will be defined as the best response at any time point per PERCIST. The metabolic response rate (complete + partial metabolic response) will be ascertained and compared between subjects treated with 17b-estradiol harboring amplified/mutant ESR1 and wild-type ESR1.
Adverse event profiles | 12 months
  The number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Mary Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No